CLINICAL TRIAL: NCT01906242
Title: Hygiene Protocols for Cleaning Complete Dentures
Brief Title: Hygiene Protocol of Complete Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: PPGO016
Record Dates: First submitted 2013-05-03; First posted 2013-07-24 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Denture Hygiene Protocol
MeSH Terms: interventions — Water; Sodium Hypochlorite; Sodium Bicarbonate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water (Placebo Comparator): Patients' dentures are treated with water (placebo) once a week for 10 min.
  Interventions: Other: water
- sodium hypochlorite (Active Comparator): Patients' dentures are treated with a solution of sodium hypochlorite 0.5% once per week for 10 min
  Interventions: Other: sodium hypochlorite
- 0.5% chlorhexidine (Active Comparator): Patients' dentures are treated with 0.5% chlorhexidine once a week for 10 min.
  Interventions: Other: chlorhexidine
- 0.12% sodium bicarbonate (Active Comparator): Patients' dentures are treated with sodium bicarbonate 0.12% once a week for 10 min.
  Interventions: Other: sodium bicarbonate

INTERVENTIONS:
Other: water
  Other Names: placebo
  Arms: Water
Other: sodium hypochlorite
  Arms: sodium hypochlorite
Other: sodium bicarbonate
  Arms: 0.12% sodium bicarbonate
Other: chlorhexidine
  Arms: 0.5% chlorhexidine

SUMMARY:
Adequate denture hygiene is important to patient's oral health maintenance in particular because of Candida albicans, responsible for the development of denture stomatitis. The aim of this study is to conduct a randomized controlled trial seeking for the best hygiene protocols to be used in removable denture wearers. The null hypothesis tested is that there will be no difference among the denture hygiene protocols tested.

ELIGIBILITY:
Inclusion Criteria:

* Complete denture wearer
* healthy
* ability to comply with the experimental protocol

Exclusion Criteria:

* Candidiasis (thrush)
* use of antifungals, antibiotics or mouthwashes in the prior 3 months
* limited motor activity
* unhealthy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Amount of biofilm formed on the denture | 14 days
  Biofilm will be measured on the denture using photographs and microbial counts (baseline and after 14 days of use of one of the four hygiene protocols) after using one of the tested denture hygiene protocols. The four tested protocols (NaOCl, chlorhexidine, sodium bicarbonate, water) will be compared to see which one leads to a better hygiene of the denture.

SECONDARY OUTCOMES:
Odor | 14 days
  Patients will be asked about the odor of the solution used to soak dentures through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Pereira-Cenci, PhD, Principal Investigator — Federal University of Pelotas; Maximiliano S Cenci, PhD, Study Chair — Federal University of Pelotas
Locations (1):
- School of Dentistry, Pelotas, Rio Grande do Sul, Brazil